CLINICAL TRIAL: NCT03112980
Title: Randomized, Multi-Center, Event-Driven Trial of TAVI Versus SAVR in Patients With Symptomatic Severe Aortic Valve Stenosis and Intermediate Risk of Mortality, as Assessed by STS-Score - DEDICATE
Brief Title: Randomized Trial of TAVI vs. SAVR in Patients With Severe Aortic Valve Stenosis at Low to Intermediate Risk of Mortality
Acronym: DEDICATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other); The German Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEDICATE; DEDICATE - DZHK 6 (Other: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK))
Record Dates: First submitted 2017-03-21; First posted 2017-04-13 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Valve Stenosis; Transcatheter Aortic Valve Replacement; Surgical aortic valve replacement; Low to intermediate operative risk
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcatheter aortic valve implantation (Experimental): Transcatheter aortic valve implantation (TAVI) using the most appropriate CE (Conformité Européene)-marked device available, with a minimum demand of experience of 30 implanted devices/type per center.
  Interventions: Device: Transcatheter aortic valve implantation
- Surgical aortic valve replacement (Active Comparator): Surgical aortic valve replacement (SAVR) with free choice of surgical bioprosthesis and free choice of surgical access according to the surgeon's preference.
  Interventions: Procedure: Surgical aortic valve replacement

INTERVENTIONS:
Device: Transcatheter aortic valve implantation — (TAVI)
  Arms: Transcatheter aortic valve implantation
Procedure: Surgical aortic valve replacement — (SAVR)
  Arms: Surgical aortic valve replacement

SUMMARY:
Randomized controlled, multi-center trial randomizing patients with symptomatic severe aortic stenosis at low to intermediate operative risk of mortality in a 1:1 fashion to transcatheter aortic valve implantation (TAVI) or surgical aortic valve replacement (SAVR) to test, whether TAVI is non-inferior to SAVR, as measured by all-cause mortality or stroke after 1 and 5 years.

DETAILED DESCRIPTION:
A paradigm-shift towards performing TAVI in intermediate- and low-risk patients has already begun, as procedural results of TAVI have improved significantly within the past years. Nevertheless, a prospective and independent comparison of surgical (SAVR) and interventional (TAVI) valve therapy in patients considered at low to intermediate risk that covers an "all-comers" patient population and multiple devices has not yet been performed.

The DEDICATE-trial is designed as a prospectively randomized (1:1), multi-center, comparator-controlled interventional trial to investigate whether transcatheter aortic valve implantation (TAVI) is non-inferior - as measured by all-cause mortality or stroke after 1 and 5 years - compared to surgical aortic valve replacement (SAVR) in the treatment of patients with symptomatic severe aortic stenosis at low to intermediate operative risk of mortality, as assessed by the local Heart Team.

ELIGIBILITY:
Inclusion Criteria:

1. Heart team consensus that TAVI and SAVR are both medically justified and advisable based on:

   1. Degenerative aortic valve stenosis with echocardiographically derived criteria:

      * Mean gradient >40 mmHg or
      * Jet velocity greater than 4.0 m/s or
      * Aortic valve area (AVA) of < 1.0 cm2 (indexed effective orifice area < 0.6cm2/m2).
   2. Patient is symptomatic from his/her aortic valve stenosis

      * New York Heart Association Functional Class ≥ II or
      * Angina pectoris or
      * Syncope.
   3. Patient is classified as low to intermediate operative risk as assessed by the local heart team according to the variables outlined in the 2017 ESC/EACTS Guidelines for the Management of valvular heart disease, taking into account cardiac and extracardiac Patient characteristics and established risk scores (e.g. STS-PROM, EuroSCORE).
   4. A transfemoral or alternative (e.g. transapical, transaortic, transaxillary) access for TAVI seems feasible. Centers should follow a "transfemoral first" strategy for the primary route of access; however, other routes of access are also allowed, as decided by local heart team consensus.
2. Patient has provided written informed consent to participate in the trial.
3. Ability of the patient to understand the patient information and to personally sign and date the informed consent to participate in the study, before performing any study related procedures.
4. The patient agrees to undergo SAVR, if randomized to control treatment.
5. The patient and the treating physician agree that the patient will return for all required post-procedure follow-up visits.
6. Patients aged 65 to 85 years.
7. Male patients or females who are postmenopausal defined as no menses for 12 months without an alternative medical cause.

Exclusion Criteria:

1. Aortic valve is a congenital unicuspid or congenital bicuspid valve, or is non-calcified
2. Untreated clinically significant coronary artery disease considered a contraindication to an isolated aortic valve procedure (TAVI or SAVR) according to heart team consensus
3. Previous cardiac surgery
4. Any percutaneous coronary intervention performed within 1 month prior to the study procedure
5. Untreated severe mitral or tricuspid regurgitation
6. Untreated severe mitral stenosis
7. Hemodynamic instability requiring inotropic support or mechanical circulatory support
8. Ischemic stroke or intracranial bleeding within 1 month
9. Severe ventricular dysfunction with left ventricular ejection fraction < 20% as measured by resting echocardiogram
10. Hypertrophic obstructive cardiomyopathy or severe basal septal hypertrophy with outflow gradient
11. Echocardiographic evidence of an intracardiac mass, thrombus, vegetation or endocarditis
12. Any other condition considered a contraindication for an isolated aortic valve procedure
13. Symptomatic carotid or vertebral artery disease
14. Expected life expectancy < 12 months due to associated non-cardiac comorbidities
15. Currently participating in another investigational drug or device trial

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1414 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from stroke or death | within 5 years after randomization
  (Efficacy endpoint)
Freedom from stroke or death | within 1 year after randomization
  (Safety endpoint)

SECONDARY OUTCOMES:
Freedom from stroke or death | Five years after last patient in
  will be assessed at every study visit and compared between TAVI and SAVR groups
Overall survival | Five years after last patient in
  will be assessed at every study visit and compared between TAVI and SAVR groups
Freedom from cardiovascular mortality | Five years after last patient in
  will be assessed at every study visit and compared between TAVI and SAVR groups
Freedom from the composite of all-cause mortality and stroke | Five years after last patient in
  will be assessed at every study visit and compared between TAVI and SAVR groups
Freedom from myocardial infarction | Five years after last patient in
  will be assessed at every study visit and compared between TAVI and SAVR groups
Freedom from stroke | Five years after last patient in
  will be assessed at every study visit and compared between TAVI and SAVR groups
Freedom from major or life-threatening / disabling bleeding | Five years after last patient in
  will be assessed at every study visit and compared between TAVI and SAVR groups
Freedom from acute kidney injury | Five years after last patient in
  will be assessed at every study visit and compared between TAVI and SAVR groups
Freedom from vascular access site and access-related complications | Five years after last patient in
  will be assessed at every study visit and compared between TAVI and SAVR groups
Freedom from conduction disturbances and arrhythmias, need for permanent pacemaker implantation | Five years after last patient in
  will be assessed at every study visit and compared between TAVI and SAVR groups
Freedom from residual aortic regurgitation ≥ moderate | Five years after last patient in
  will be assessed at every study visit and compared between TAVI and SAVR groups
Composite device success | Five years after last patient in
  Number of participants with freedom from procedural mortality and correct positioning of a single transcatheter heart valve (THV) in the proper position with intended performance (no prosthesis- patient mismatch and mean aortic valve gradient <20 mmHg or peak velocity <3 m/s, AND no moderate or severe prosthetic valve regurgitation)
Composite early safety | within first 30 days after procedure
  Number of participants dying and/or number of participants with stroke (disabling and non-disabling), and/or life-threatening bleeding and/or acute kidney injury stages 2/3 and/or coronary artery obstruction requiring Intervention and/or major vascular complication and/or valve-related dysfunction requiring repeat procedure.
Composite clinical efficacy | within first 30 days after procedure
  Number or participants dying and/or number of participants with stroke (disabling and non-disabling) and/or rehospitalisation for worsening heart failure or valve-related symptoms and/or New York Heart Association functional class (NYHA) III or IV and/or valve-related dysfunction (mean aortic valve gradient >20 mmHg, effective orifice area (EOA) <0.9-1.1 cm2 and/or Doppler Velocity Index (DVI) <0. 35 m/s, AND/OR moderate or severe prosthetic valve regurgitation)
Freedom from prosthetic valve dysfunction | Five years after last patient in
  will be assessed at every study visit and compared between TAVI and SAVR groups
Freedom from prosthetic aortic valve endocarditis | Five years after last patient in
  will be assessed at every study visit and compared between TAVI and SAVR groups
Freedom from the composite time-related valve safety | Five years after last patient in
  Number of participants with structural valve deterioration (including repeat procedures, prosthetic valve endocarditis and/or thrombosis) and/or number of participants with thromboembolic events (stroke) and/or Valve Academic Research Consortium (VARC-2) bleeding (unless clearly unrelated to valve therapy).
Quality of life measures | Five years after last patient in
  Number of participants with reduced quality of life measures after valve replacement as compared to baseline levels prior to valve-replacement, assessed using EuroQol five dimensions (EQ-5D) questionnaire and/or Barthel Index and/or center for epidemiologic studies depression (CES-D) Scale.
Health economic analysis | Five years after last patient in
  Incremental cost-effectiveness of TAVI compared to surgical valve replacement, by using quality adjusted life years (QALYs).
Number of (re) hospitalisations | Five years after last patient in
  Number rehospitalisations of all participants. Length of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Blankenberg, MD, Principal Investigator — Universitäres Herz- und Gefäßzentrum Hamburg (UHZ), Germany; Jochen Cremer, MD, Principal Investigator — Universitätsklinikum Schleswig-Holstein, Germany
Locations (43):
- Germany (43):
  - Uniklinik Rheinisch-Westfälische Technische Hochschule Aachen, Aachen
  - Universitäts-Herzzentrum Freiburg-Bad Krozingen, Bad Krozingen
  - Kerckhoff-Klinik Bad Nauheim, Bad Nauheim
  - Herz- und Gefässklinik Bad Neustadt/Saale, Bad Neustadt an der Saale
  - Herz- und Diabeteszentrum NRW Bad Oeynhausen, Bad Oeynhausen
  - Charité Universitätsmedizin Berlin (Campus Benjamin-Franklin), Berlin
  - Charité Universitätsmedizin Berlin (Campus Mitte), Berlin
  - Charité Universitätsmedizin Berlin (Campus Virchow), Berlin
  - Deutsches Herzzentrum Berlin, Berlin
  - Vivantes Friedrichshain, Berlin
  - Vivantes Humboldt Kliniken, Berlin
  - Vivantes Klinikum am Urban, Berlin
  - Vivantes Neukölln, Berlin
  - Immanuel Klinikum Bernau, Bernau
  - Kliniken der Ruhr-Universität Bochum, Bochum
  - Medizinische Hochschule Brandenburg Theodor Fontane, Brandenburg
  - Herzzentrum der Uniklinik Köln, Cologne
  - Herzzentrum Dresden an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Klinikum für Kardiologie und Angiologie am Westdeutschen Herz- und Gefäßzentrum, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitäts-Herzzentrum Freiburg-Bad Krozingen, Freiburg im Breisgau
  - Universitätsklinikum Giessen und Marburg, Giessen
  - Universitätsklinikum Göttingen, Göttingen
  - Universitätsmedizin Greifswald / Klinikum Karlsburg, Greifswald / Karlsburg
  - Universitätsklinikum Halle (Saale), Halle
  - Universitäres Herz- und Gefäßzentrum Hamburg (UHZ), Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Bundeswehrzentralkrankenhaus Koblenz, Koblenz
  - Deutsches Herzzentrum Leipzig, Leipzig
  - Universitäres Herzzentrum Lübeck, Lübeck
  - Otto-von Guericke-Universität Magdeburg, Magdeburg
  - Universitätsmedizin Mainz, Mainz
  - Deutsches Herzzentrum München, München
  - LMU Klinikum der Universität München, München
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Regensburg, Regensburg
  - Robert Bosch Krankenhaus, Stuttgart
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seiffert M, Vonthein R, Baumgartner H, Borger MA, Choi YH, Falk V, Frey N, Hagendorff A, Hagl C, Hamm C, Konig IR, Landmesser U, Massberg S, Reichenspurner H, Thiele H, Twerenbold R, Vens M, Walther T, Ziegler A, Cremer J, Blankenberg S. Transcatheter aortic valve implantation versus surgical aortic valve replacement in patients at low to intermediate surgical risk: rationale and design of the randomised DEDICATE Trial. EuroIntervention. 2023 Oct 23;19(8):652-658. doi: 10.4244/EIJ-D-23-00232. PMID 37655862
- [Background] Blankenberg S, Seiffert M, Vonthein R, Baumgartner H, Bleiziffer S, Borger MA, Choi YH, Clemmensen P, Cremer J, Czerny M, Diercks N, Eitel I, Ensminger S, Frank D, Frey N, Hagendorff A, Hagl C, Hamm C, Kappert U, Karck M, Kim WK, Konig IR, Krane M, Landmesser U, Linke A, Maier LS, Massberg S, Neumann FJ, Reichenspurner H, Rudolph TK, Schmid C, Thiele H, Twerenbold R, Walther T, Westermann D, Xhepa E, Ziegler A, Falk V; DEDICATE-DZHK6 Trial Investigators. Transcatheter or Surgical Treatment of Aortic-Valve Stenosis. N Engl J Med. 2024 May 2;390(17):1572-1583. doi: 10.1056/NEJMoa2400685. Epub 2024 Apr 8. PMID 38588025